CLINICAL TRIAL: NCT07043712
Title: Human Pulse Consumption, the Microbiome, and Meal Satiety
Brief Title: Effects of Pulse Consumption, Gut Microbiome, and Appetite in Healthy Participants
Acronym: PULSE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Katherene Anguah, Associate Professor, Nutrition and Exercise Physiology, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2066363
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-06

CONDITIONS: Microbial Colonization; Metabolic Syndrome
Keywords: overweight; satiety; SCFA; pulses
MeSH Terms: conditions — Communicable Diseases; Metabolic Syndrome; Overweight

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the high pulse diet or no pulse diet.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High pulse consumption (Experimental): Subjects are provided a high pulse diet for 4-weeks. Tests include: blood biochemistries, a meal tolerance test, body composition measured via DEXA, surveys, fecal sample
  Interventions: Dietary Supplement: High pulse consumption
- No pulse consumption (No Intervention): Subjects are provided a diet that has no pulses for 4-weeks. Tests include: blood biochemistries, a meal tolerance test, body composition measured via DEXA, surveys, fecal sample

INTERVENTIONS:
Dietary Supplement: High pulse consumption — Subjects are provided a high pulse diet for 4 weeks.collection, and anthropometrics measured.
  Arms: High pulse consumption

SUMMARY:
The purpose of the study is to investigate the effects of pulse consumption versus no pulse consumption on the gut microbiome, meal satiety, and short-chain fatty acid metabolomics.

DETAILED DESCRIPTION:
1. Investigate the acute and chronic effects of pulse consumption on the microbiome and plasma SCFA metabolomics in overweight subjects fed a high pulse (n=22) diet versus a no pulse containing diet (n=22).
2. Furthermore, we will quantitate the rate of production of plasma SCFA, markers of satiety (PYY, GLP-1 and ghrelin), blood lipids, and carbohydrate (CHO) metabolism (glucose levels and oxidation) during a standardized meal to determine the effects of consuming pulses on appetite and satiety after acute and chronic dietary consumption.
3. We will conduct subjective appetite assessments to investigate appetite control over the short- and long-term.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (premenopausal only)
* Age 20-55y (we will attempt to start baseline testing at the same time of the menstrual cycle (luteal) for the women
* BMI ≥25 or ≤40 kg/m2 (most at risk for metabolic abnormalities and will benefit from a pulse intervention-2/3 of Americans are overweight or obese)
* Weight stable (no fluctuations in body weight of greater than 4 kg in the last 3 months)
* Willing to consume a research diet
* Willing to provide blood and fecal samples
* Sedentary to low active physical activity status (less than 7200 steps per day)
* Stably treated with statin drugs, anti-hypertensives, and anti-depressants. These are acceptable as long as the drug category does not alter appetite, body weight, or the microbiome (if known)
* Pre-diabetes acceptable (glucose <125 mg/dL or HbA1c < 6.5%)
* At least one characteristic of the metabolic syndrome (but not diabetic)

  1. A large waistline: 35 inches or more for women 40 inches or more for men
  2. High triglycerides: 150 mg/dL or higher
  3. Low HDLc level: <50 mg/dL for women <40 mg/dL for men
  4. High blood pressure ≥130/85 mmHg
  5. Fasting blood sugar ≥100 mg/dL - Pre-diabetes acceptable (glucose <125 mg/dL or HbA1c <6.5%) -

Exclusion Criteria:

* Pregnant or lactating
* Postmenopausal (evidence suggests an interplay between the gut microbiome)
* BMI of <25 or >40 kg/m2
* Use of medications that affect the gut microbiome (e.g. antibiotics)
* Taking medications known to affect appetite (e.g., phentermine) or gastrointestinal function (e.g., metformin)
* On a special diet or undergoing weight loss, vegetarian, or other restricted dietary patterns
* Ad libitum intake of fiber above 25g/day (mean intake in the US population is 17g/day) and < 10g/d
* History of disease (example colon cancer, HIV, cardiovascular disease, psychiatric disorders, etc.)
* Use of tobacco products

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
gut microbial change | baseline to 4 weeks
  assessed via 16s rRNA gene sequencing from fecal samples collection
Change in appetite hormones | baseline to 4 weeks
  GLP-1 measurement in plasma samples

SECONDARY OUTCOMES:
cardiometabolic risk factors | baseline to 4 weeks
  total cholesterol,
Change in subjective appetite | baseline to 4 weeks
  Subjective fullness measured via 100 mm visual analogue scale
short chain fatty acid metabolomics | baseline to 4 weeks
  plasma short chain fatty acids
Body composition | baseline to 4 weeks
  Assessed via DEXA during each of two meal test visits

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No